CLINICAL TRIAL: NCT03827421
Title: Transcranius : Junior Emergency Physician Learning Curve to Perform Transcranial Doppler on Brain-damage Patients
Brief Title: Junior Emergency Physician Learning Curve to Perform Transcranial Doppler on Brain-damage Patients
Acronym: Transcranius
Status: Terminated | Type: Observational
Why Stopped: Organizational reasons and lack of enrollment
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC18.211; 2018-A02346-49 (Other: IDRCB)
Record Dates: First submitted 2018-12-14; First posted 2019-02-01 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Brain Damage
Keywords: transcranial doppler; learning curve; emergency; traumatic brain injury
MeSH Terms: conditions — Brain Injuries; Emergencies; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Transcranial Doppler is a noninvasive tool. Using velocity measurements and pulsatility index it allows the evaluation of cerebral haemodynamics. In patients presenting brain injury cerebral perfusion may be impaired. Indirect cerebral blood flow can be monitored and risk of neurological worsening can be detected using transcranial Doppler. Education and performance of emergency physicians must be evaluated on brain-injured patients because this tool is operator dependent. The main objective of this study is to estimate the average number of exams required to learn transcranial Doppler within junior emergency physicians with the achievement of their learning curve. We will perform a prospective, monocentric, observational study within the neurosurgical resuscitation department of Grenoble Alpes University Hospital.

DETAILED DESCRIPTION:
The transcranial dopplers will be carry out on 75 brain-damaged patients by 13 emergency residents physicians after a theoretical and practical training. They will be evaluated by 8 experts. The primary endpoint will be the mean number of transcranial dopplers required to have an excellent concordance between resident and expert. The concordance between the Doppler findings of the resident and the expert would exceed 0.8 before 30 examinations. The learning curve assessed on the duration necessary to acquire good quality data should decrease rapidly with the repetition of the examinations. Validating the transcranial Doppler learning curve for junior emergency physician would allow them to perform this exam safely and efficiently. Transcranial Doppler may be easy and fast to learn but the persistence of its competency over time should be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients : ≥ 18 year and older
* Hospitalized in the neurosurgical resuscitation or intensive care unit
* Brain - damaged patients

Exclusion Criteria:

* Any craniotemporal lesion impeding satisfactory TDC examination : no transtemporal doppler window, patient with craniectomy.
* Patient with meningo-encephalitis
* Patient with cerebral vasculitis
* Patient without health insurance coverage
* Patient subject to a legal protection measure
* Pregnant woman , parturient or nursing

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Brain-damaged patients hospitalized in neurosurgical resuscitation or intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The mean number of transcranial doppler required to reach a kappa over 0,8 between the conclusions of the resident and expert. | 3 months
  Learning curve

SECONDARY OUTCOMES:
Duration in seconds for the junior to achieve the transcranial doppler | 3 months
  Time between the beginning of the exam (ultrasound probe caring) to the velocities and pulsatility index measurements
Analysis of the spectral envelope quality | 3 months
  analysis of the plot of spectral envelope: good or bad
Analysis of the evolution of the estimated difficulty of transcranial doppler realization | 3 months
  evaluation of the difficulty of transcranial doppler realization: easy or difficult
Analysis of the failure to perform the transcranial doppler | 10 minutes
  number of failures to perform the transcranial doppler after 10 minutes
Analysis of the diastolic velocities and pulsatility index concordance between junior and expert | 3 months
  number of examen required for junior velocities measurement to reach those of the expert

CONTACTS AND LOCATIONS:
Overall Officials: Batistin MARTINON, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, Auvergne Rhonalpes, France

IPD SHARING:
Plan to Share IPD: No